CLINICAL TRIAL: NCT01137058
Title: Clinical Efficacy of Ubiquitous Healthcare System for Elderly Patients With Type 2 Diabetes Mellitus
Brief Title: Ubiquitous Healthcare for Elderly Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SNUBH_UH1
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- U-healthcare (Experimental): glucose meter and U-healthcare
  Interventions: Device: U-healthcare service
- SMBG group (Active Comparator): Diabetic patients who do self monitoring of blood glucose only were categorized into self monitoring of blood glucose (SMBG) group.
  Interventions: Device: SMBG group
- control (No Intervention): conventional treatment

INTERVENTIONS:
Device: U-healthcare service — Public switched telephone network (PSTN)-connected glucometer with U-healthcare system.
  Other Names: U-healthcare group
  Arms: U-healthcare
Device: SMBG group — Glucose control with self monitoring of blood glucose.
  Arms: SMBG group

SUMMARY:
Ubiquitous healthcare service for elderly patients with type 2 diabetes provides real-time glycemic monitoring and glucose control implemented by clinical decision support system (CDSS) using wire and wireless communication and information technology.

To evaluate the clinical efficacy of this system, researchers plan to compare the improvement of glycemic control, self-management, and quality of life among three study groups: control, self glucose monitoring, and U-healthcare group.

DETAILED DESCRIPTION:
Recently, the application of internet-based glucose control system showed better long term glucose control compared to the conventional treatment. This study has become the foundation of web-based methodology in the glucose control. In addition, the combined application of mobile device and web-based monitoring system for chronic diseases showed improvement in various metabolic parameters in obese patients with diabetes and hypertension.

Thus, the application of U-healthcare based on advanced information technology would be helpful in the diabetes management. We plan to provide an individualized U-healthcare service using advanced information technology that enables more effective glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* age: 60 ~ 85 yrs
* HbA1c: 6.5%-11.0%
* duration of diabetes: less than 30 years
* BMI: 20-35

Exclusion Criteria:

* systemic corticosteroid administered within previous 6 months
* history of myocardial ischemia
* Heart failure, NYHA Class II-IV
* Thyroid disease with abnormal TFT
* Anti-obesity drugs or slimming products within previous 3 months

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Target goal of HbA1c (< 7.0%) without hypoglycemia | 24 weeks
  Percent of patients who reach target goal of HbA1c (< 7.0%) without hypoglycemia

SECONDARY OUTCOMES:
quality of life | 24 weeks
amount of exercise | 24 weeks
Body mass index (BMI) changes | Body mass index
  Comparison of body mass index changes among control, self monitoring of blood glucose (SMBG) and ubiquitous healthcare groups

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, MPH, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

REFERENCES:
- [Derived] Lim S, Kang SM, Kim KM, Moon JH, Choi SH, Hwang H, Jung HS, Park KS, Ryu JO, Jang HC. Multifactorial intervention in diabetes care using real-time monitoring and tailored feedback in type 2 diabetes. Acta Diabetol. 2016 Apr;53(2):189-98. doi: 10.1007/s00592-015-0754-8. Epub 2015 May 5. PMID 25936739
- [Derived] Lim S, Kang SM, Shin H, Lee HJ, Won Yoon J, Yu SH, Kim SY, Yoo SY, Jung HS, Park KS, Ryu JO, Jang HC. Improved glycemic control without hypoglycemia in elderly diabetic patients using the ubiquitous healthcare service, a new medical information system. Diabetes Care. 2011 Feb;34(2):308-13. doi: 10.2337/dc10-1447. PMID 21270188